CLINICAL TRIAL: NCT01520337
Title: Polyp Detection Rate After Single Oral Dose of Methylene Blue MMX Modified Release Tablets Administered to Subjects Undergoing Outpatients Colonoscopy
Status: Completed | Type: Observational
Sponsor: Cosmo Technologies Ltd (Industry)
Responsible Party: Sponsor
Organization: CosmoTech (Unknown)
Other Study IDs: CB-17-01/05; 2011-005694-23 (EudraCT Number)
Record Dates: First submitted 2012-01-25; First posted 2012-01-27 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Polyp and Adenoma Detection During Colonoscopy
MeSH Terms: conditions — Polyps

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — mucosal biopsy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients undergoing outpatient colonoscopy
  Interventions: Device: oral tablet dye for detection of polyps during colonoscopy

INTERVENTIONS:
Device: oral tablet dye for detection of polyps during colonoscopy — oral tablet dye for improved detection of

SUMMARY:
Polyp detection rate in colonoscopy following oral administration of MMX methylene blue tablets

DETAILED DESCRIPTION:
Polyp detection rate in colonoscopy following oral administration of methylene blue MMX modified release tablets in subjects undergoing colonoscopy as outpatients.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for screening or surveillance colonoscopy. Written informed consent.Practising reliable contraception or sterile.Ability to understand and comply with the protocol.

Exclusion Criteria:

* Pregnancy or lactation known or suspected hypersensitivity GI obstruction or perforation serious cardiovascular, renal or hepatic disease. reduced prothrombin time,elevated serum creatinine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for screening or surveillance colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Polyp and adenoma detection rate | 1 day